CLINICAL TRIAL: NCT03419130
Title: A Phase II Study of Radiation Therapy and Pembrolizumab in Patients With Localized Urothelial Bladder Cancer That Are Ineligible or Refusing Chemotherapy
Brief Title: Radiation Therapy and Pembrolizumab in Treating Patients With Localized Urothelial Bladder Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn prior to patient enrollment
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17522; NCI-2017-02196 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-22452; 17522 (Other: UCSF Medical Center-Mount Zion)
Record Dates: First submitted 2017-12-08; First posted 2018-02-01 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Infiltrating Bladder Urothelial Carcinoma; Stage II Bladder Urothelial Carcinoma AJCC v6 and v7; Stage III Bladder Urothelial Carcinoma AJCC v6 and v7
MeSH Terms: interventions — Radiation Dose Hypofractionation; pembrolizumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (pembrolizumab, hypofractionated RT) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 13 courses in the absence of disease progression or unacceptable toxicity. Patients also receive hypofractionated RT over 5 fractions for 14 days.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab
- Cohort II (pembrolizumab, conventionally fractionated RT) (Experimental): Patients receive pembrolizumab as in Cohort I. Patients also receive conventionally fractionated RT over 30 fractions for 52 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated RT
  Other Names: Hypofractionated Radiotherapy; hypofractionation
  Arms: Cohort I (pembrolizumab, hypofractionated RT)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Radiation: Radiation Therapy — Undergo conventionally fractionated RT
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Cohort II (pembrolizumab, conventionally fractionated RT)

SUMMARY:
This randomized phase II trial studies how well radiation therapy and pembrolizumab work in treating patients with urothelial bladder cancer that is restricted to the site of origin, without evidence of spread. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Giving radiation therapy and pembrolizumab may work better in treating urothelial bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximally tolerated doses of hypofractionated and conventionally fractionated radiation therapy in combination with pembrolizumab and to generate an estimate of the efficacy of this regimen. (Safety Lead-in) II. To estimate the clinical complete response (CR) rate of the primary irradiated tumor in patients receiving radiotherapy and pembrolizumab. (Dose Expansion Cohort)

SECONDARY OBJECTIVES:

I. To estimate the local control rate at 6 and 12 months in each study arm. II. To estimate the distant metastases free survival at 6 and 12 months in each study arm.

III. To estimate progression free survival at 6 and 12 months in each study arm.

IV. To estimate disease-specific survival at 6 and 12 months in each study arm. V. To determine the safety of combining radiotherapy with pembrolizumab in each study arm in the dose expansion phase.

TERTIARY OBJECTIVES:

I. To assess peripheral and tumor-based biomarkers of response and resistance. II. To define the treatment-induced effects on circulating immune cells. III. To explore the remodeling of circulating T cell repertoire.

OUTLINE: Patients are randomized to 1 of 2 cohorts.

COHORT I: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Treatment repeats every 3 weeks for up to 13 courses in the absence of disease progression or unacceptable toxicity. Patients also receive hypofractionated radiation therapy (RT) over 5 fractions for 14 days.

COHORT II: Patients receive pembrolizumab as in Cohort I. Patients also receive conventionally fractionated RT over 30 fractions for 52 weeks.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Localized, muscle invasive urothelial carcinoma (T2-4, N0-1, M0) (mixed histology acceptable) ineligible for cystectomy
* Patients must not be suitable for concurrent cisplatin as determined by the following:

  * Creatinine clearance less than 60ml/min; glomerular filtration rate (GFR) should be assessed by calculation from serum/plasma creatinine (Cockcroft-Gault formula)
  * Common Terminology Criteria for Adverse Events (CTCAE) grade (Gr) >= 2 hearing loss
  * CTCAE Gr >= 2 neuropathy
* Patients must not be suitable for fluorouracil (5FU)/mitomycin chemotherapy
* Subjects with not meeting the above criteria are still eligible provided the patient declines concurrent chemotherapy with radiation, after specific informed consent describing the known benefits of adding chemotherapy to the definitive bladder radiation regimen; the reason for declining must be documented
* Life expectancy of at least 3 months or greater
* Be willing and able to provide written informed consent/assent for the trial
* Be willing to provide tissue from a newly obtained transurethral resection of bladder tumor (TURBT) or biopsy of a tumor lesion; newly-obtained is defined as a specimen obtained up to 8 weeks (56 days) prior to initiation of treatment on say 1; subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the sponsor
* Have a performance status of 0 - 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) >= 1,500 /mcL, performed within 28 days of treatment initiation
* Platelets >= 100,000 / mcL, performed within 28 days of treatment initiation
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment), performed within 28 days of treatment initiation
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or creatinine clearance [CrCl]) >= 30 mL/min for subject with creatinine levels > 1.5 X institutional ULN, performed within 28 days of treatment initiation
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN, performed within 28 days of treatment initiation
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X ULN, performed within 28 days of treatment initiation
* Albumin >= 2.5 mg/dL, performed within 28 days of treatment initiation
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants, performed within 28 days of treatment initiation
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants, performed within 28 days of treatment initiation
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 120 days after the last dose of study medication

  * Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Male subjects of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy

  * Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

Exclusion Criteria:

* Non-muscle invasive, localized bladder cancer (Tis, Ta, T1)
* Presence of distant metastatic disease or disease not amenable to radiation treatment
* Prior radiation treatment to the pelvis
* Prior cystectomy
* Is currently participating and receiving study therapy, or has participated in a study of an investigational agent and received study therapy, or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has a known history of active tuberculosis (TB) (Mycobacterium tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Prior systemic chemotherapy for bladder cancer; prior intravesical chemotherapy for the treatment of non-muscle invasive urothelial bladder cancer (UBC) is allowed
* Upper tract urothelial carcinoma
* Has had prior chemotherapy or targeted small molecule therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known distant metastases; clinically involved pelvic nodes (N1-N3) are allowed
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment; topical and inhaled corticosteroids are allowed
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject?s participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Has known active hepatitis B (e.g., hepatitis B virus surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)

  * Patients with past hepatitis B virus (HBV) infection or resolved HBV infection, defined as the presence of hepatitis B core antibody (HBc Ab) and absence of hepatitis B surface antigen (HBsAg) are eligible; HBV deoxyribonucleic acid (DNA) must be obtained in these patients prior to day 1 of therapy, but detection of HBV DNA in these patients will not exclude study participation
  * Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans)
* Has a history of (non-infectious) pneumonitis that required steroids, or has current pneumonitis
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-18 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
cCR rate (expansion cohort) | Up to 24 months
  A complete response will be defined as the absence of visible tumor endoscopically (cystoscopically) and the absence of histologic evidence of disease if a biopsy is performed.
Clinical complete response (cCR) rate (safety lead-in) | At 12 weeks
  A cCR rate will be defined at week 12 after the initiation of study therapy as no residual muscle-invasive disease (=< T1) on cystoscopy. This rate will be summarized using descriptive statistics. The point estimate of cCR rate will be obtained with its 95% confidence intervals.
Incidence of adverse events evaluated according to Common Terminology Criteria for Adverse Events version 4.3 (safety lead-in) | Up to 12 weeks
  Safety will be summarized using descriptive statistics.

SECONDARY OUTCOMES:
Disease specific survival (DSS) | At 6 months
  DSS will be compared between two arms by the stratified log-rank test.
Distant metastasis free survival (DMFS) | At 6 months
  DMFS will be compared between two arms by the stratified log-rank test.
DMFS | At 12 months
  DMFS will be compared between two arms by the stratified log-rank test.
DSS | At 12 months
  DSS will be compared between two arms by the stratified log-rank test.
Incidence of adverse events evaluated according to CTCAE version 4.3 | Up to 24 months
  Safety and tolerability in all phases will be summarized by maximum toxicity grade for each study arm. The toxicity grade for laboratory data will be calculated using CTCAE version (v)4.3 and the lab data will be summarized according to the subjects baseline grade and maximum grade for each course of therapy. All treatment related adverse events will be graded using National Cancer Institute CTCAE v4.3 and will be recorded and listed.
Local control (LC) rate | Up to 12 months
  The point estimate of LC rate will be summarized descriptively at each specified time point from 6-12 months after therapy using descriptive statistics with 95% confidence interval for each arm.
Progression Free Survival (PFS) | At 12 months
  PFS will be compared between two arms by the stratified log-rank test.
Progression-free survival (PFS) | At 6 months
  PFS will be compared between two arms by the stratified log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Terence Friedlander, Principal Investigator — UCSF Medical Center-Mount Zion
Locations (1):
- UCSF Medical Center-Mount Zion, San Francisco, California, United States